CLINICAL TRIAL: NCT06507202
Title: Comparison of Remimazolam Versus Propofol-based General Anesthesia on Postoperative Quality of Recovery in Patients Undergoing Ambulatory Upper Airway Surgery: a Randomized Controlled Trial
Brief Title: Comparison of Remimazolam and Propofol for Recovery of Ambulatory Upper Airway Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chung-Ang University Gwangmyeong Hospital (Other)
Responsible Party: Principal Investigator, Se-Hee Min, Assistant professor, Chung-Ang University Gwangmyeong Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2311123132
Record Dates: First submitted 2024-01-18; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Laryngeal Disease; Pharyngeal Diseases; Oral Cavity Disease; Nasal Disease
Keywords: remimazolam; upper airway surgery; ambulatory surgery
MeSH Terms: conditions — Laryngeal Diseases; Pharyngeal Diseases; Mouth Diseases; Nose Diseases | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): General anesthesia is induced by continuously injecting remimazolam (6 mg/kg/h) and remifentanil (2-6 ng/ml, target concentration controlled infusion) through an infusion pump. Afterwards, when the patient loses consciousness, rocuronium 0.6 mg/kg is injected for endotracheal intubation, and anesthesia is maintained with remimazolam (1-2 mg/kg/hr) and remifentanil after endotracheal intubation. When the surgery is completed, all anesthetic drugs being administered are stopped, and general anesthesia is terminated with flumazenil and sugammadex.
  Interventions: Drug: Remimazolam
- Propofol group (Active Comparator): General anesthesia is induced by continuously injecting propofol (2-6 mg/ml, target concentration controlled injection) and remifentanil (2-6 ng/ml, target concentration controlled injection) using a TCI infusion pump. Afterwards, when the patient loses consciousness, rocuronium 0.6mg/kg is injected for endotracheal intubation, and anesthesia is maintained with propofol and remifentanil after endotracheal intubation. When the surgery is completed, all anesthetic drugs being administered are stopped, and general anesthesia is terminated through sugammadex.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — General anesthesia is induced and maintained by continuous infusion of remimazolam and remifentanil, and recovered with flumazenil.
  Other Names: Byfavo
  Arms: Remimazolam group
Drug: Propofol — General anesthesia is induced and maintained by continuous infusion of propofol and remifentanil.
  Other Names: Fresofol
  Arms: Propofol group

SUMMARY:
The purpose of this study is to compare the effects of remimazolam and propofol on postoperative recovery time, complications, and safety in patients undergoing ambulatory upper airway surgery under general anesthesia.

DETAILED DESCRIPTION:
Patients scheduled for ambulatory upper airway (including nasal cavity, oral cavity, pharynx, larynx) surgery and who agree to participate in the study will be randomly assigned to the Remimazolam group and the Propofol group. In the Remimazolam group, general anesthesia is induced and maintained by continuous infusion of remimazolam and remifentanil. Once the surgery is completed, general anesthesia is recovered with flumazenil. In the Propofol group, general anesthesia is induced and maintained by continuous infusion of propofol and remifentanil using a target concentration controlled infusion method. In both groups, rocuronium is used for neuromuscular blokade, and sugammadex is used for reversal of neuromuscular blockade.

When the surgery is completed, recovery time, occurrence of adverse events, and anesthesia recovery indicators are examined in 3 stages: in the operating room, while staying in the post-anesthesia care unit(PACU), and while staying in the day surgery center.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 19 or older) undergoing ambulatory upper respiratory tract (nasal cavity, oral cavity, pharynx, larynx) surgery under general anesthesia
* American Society of Anesthesiologists physical class classification I, II, and III

Exclusion Criteria:

* Patients who refused to participate in the study
* Pregnant patients
* Patients with a history of hypersensitivity to drugs or additives used during surgery
* Patients with acute narrow-angle glaucoma
* Alcohol or drug dependent patients
* Patients with Child-Pugh class C liver dysfunction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-01-22 (Estimated); Study Completion 2025-03-22 (Estimated)

PRIMARY OUTCOMES:
Fit-for-discharge time | 15 minutes after surgery
  Evaluated on a scale of 0 to 10 through the Modified Post Anesthetic Discharge Scoring System (MPADSS); a score of 9 or higher meets the discharge criteria.

SECONDARY OUTCOMES:
Time to eye opening, time to extubate, time to postanesthetic care unit (PACU) transfer | 1 minute
  Measured at operating room, using a timer from the end of surgery
postanesthetic care unit (PCAU) stay time, Day surgery center stay time | 5 minutes
  Measured from entering to exiting each units
Incidence of adverse events | 6 hours
  Including desaturation, laryngospasm, hypotension, bradycardia, hemodynamic agent administration, emergence agitation, headache, dizziness, somnolence, cough, shivering, postoperative nausea & vomiting
Postoperative pain score | 6 hours
  11-point NRS (0-10); for the worst pain
modified Observer's Alertness/Sedation Scale (MOAA/S) at PACU arrival | 30 minutes
  Evaluated on a scale of 0 to 5
modified Aldrete score at PACU arrival | 30 minutes
  Evaluated on a scale of 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hee Min, Study Chair — Chung-Ang University Gwangmyeong Hospital
Locations (1):
- ChungAng University Gwangmyeong Hospital, Gyeonggi-do, Gwangmyeon-si, South Korea

IPD SHARING:
Plan to Share IPD: No